CLINICAL TRIAL: NCT07398768
Title: A Prospective, Non-interventional, Single-Centre Study Assessing the Time Course of a Holistic Perioral Rejuvenation Procedure
Brief Title: Prospective, Non-interventional Study Assessing Perioral Rejuvenation Procedure
Status: Not yet recruiting | Type: Observational
Sponsor: Yuvell (Other)
Collaborators: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: YUV-NIS-003
Record Dates: First submitted 2026-02-02; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Perioral Wrinkles; Crow's Feet; Lip Volume Enhancement; Lip Aging
Keywords: smoker's lines; perioral wrinkles; perioral lines; hyaluronic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Saypha® Rich — Device is used as part of routine clinical care. This observational study does not assign or modify treatment; it observes outcomes associated with device use.
  Other Names: hyaluronic acid
Device: Saypha® Filler Lidocaine — Device is used as part of routine clinical care. This observational study does not assign or modify treatment; it observes outcomes associated with device use.
  Other Names: hyaluronic acid with lidocaine

SUMMARY:
The goal of this observational study is to learn how a perioral rejuvenation procedure affects perioral line severity and lip volume over time in adults undergoing routine aesthetic treatment in a single clinical center. The main questions it aims to answer are:

* What proportion of participants achieves a ≥1-point improvement from baseline on both the Lip Fullness Scale (LFS) and the Static Perioral Lines Assessment Scale (SPLAS) at Week 12?
* How do skin wrinkling/surface roughness, lip and perioral volume, and patient satisfaction change over 6 and 12 weeks?

Participants will:

* Receive a routine (non-study-mandated) holistic perioral rejuvenation procedure as decided by their treating clinician.
* Attend study visits at approximately baseline, Week 6, and Week 12.
* Undergo independent clinical assessments (assessor not involved in treatment delivery) of LFS and SPLAS.
* Have skin wrinkling and surface roughness documented by VISIA skin analysis (baseline, Week 6, Week 12).
* Have lip and perioral volume measured by VECTRA M3 volume analysis (baseline, Week 6, Week 12).
* Complete a standardized patient satisfaction questionnaire (Week 12).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older at time of treatment.
2. At least mild static perioral lines and maximum of thin lips, as assessed by the investigator.
3. Participant has a stable medical condition with no uncontrolled systemic disease.
4. Willingness to participate in the routine follow-up after 12 weeks and a signed ICF.
5. Participant already visiting the clinic for the specific treatment.

Exclusion Criteria:

1. Pregnancy and breast feeding.
2. Known impairment of blood coagulation.
3. Presence of acute infection or inflammation at the proposed injection sites.
4. Hyaluronic Acid-Filler treatment in the perioral area within the last 6 months.
5. Patients with a history of autoimmune disease or who are receiving immune therapy.
6. History of hypersensitivity to hyaluronic acid, lidocaine hydrochloride or other amidetype local anaesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the clinic for such a treatment as part of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a combined ≥ 1-point improvement in perioral line severity and lip fullness at Week 12 | Week 12
  Proportion of participants achieving a combined responder status, defined as an improvement of at least 1 point from baseline on both perioral line severity and lip fullness at Week 12, as assessed by an independent investigator not involved in treatment procedures, using the following validated photo-numeric scales:
  * Upper and lower lip fullness assessed using the Lip Fullness Scale (LFS), a validated 5-point photo-numeric rating scale ranging from Grade 1 (very thin) to Grade 5 (full), where higher scores indicate greater lip fullness. The upper and lower lips are graded separately.
  * Static perioral line severity assessed using the Static Perioral Lines Assessment Scale (SPLAS), a photo-numeric scale ranging from 1 (none) to 5 (very severe), where higher scores indicate greater severity of perioral lines.
  A participant is considered a responder only if the ≥ 1-point improvement criterion is met on both the LFS and the SPLAS simultaneously relative to baseline.

SECONDARY OUTCOMES:
Change in skin wrinkling and surface roughness of the lips and perioral region assessed by VISIA® skin analysis | Week 6, Week 12
  Change from baseline in skin wrinkling and surface roughness of the lips and perioral region, assessed at Week 6 and Week 12 using the VISIA® Skin Analysis System (Canfield).
  Skin wrinkling and surface roughness are quantified as percentage-based measurements derived from standardized, high-resolution VISIA images captured frontally and obliquely. For this outcome, values are calculated as the mean percentage from frontal images obtained at each time point.
  The outcome is expressed as the change in percentage points relative to baseline, with higher percentage values indicating improvement, corresponding to reduced skin wrinkling and smoother skin surface in the lips and perioral region.
Change in combined upper and lower lip fullness assessed by the Lip Fullness Scale (LFS) | Week 6, Week 12
  Change from baseline in upper and lower lip fullness, assessed at Week 6 and Week 12 by an independent investigator who is not involved in treatment delivery or injection procedures, using the Lip Fullness Scale (LFS).
  The LFS is a validated 5-point photo-numeric rating scale ranging from Grade 1 (very thin) to Grade 5 (full), where higher scores indicate greater lip fullness. The upper and lower lips are graded separately, and the assigned grades are recorded at each assessment time point.
  The outcome is expressed as the change in LFS score relative to baseline at each follow-up visit, reflecting changes in combined upper and lower lip volume over time.
Change in perioral line severity assessed by the Static Perioral Lines Assessment Scale (SPLAS) | Week 6, Week 12
  Change from baseline in perioral line severity, assessed at Week 6 and Week 12 by an independent investigator who is not involved in treatment delivery or injection procedures, using the Static Perioral Lines Assessment Scale (SPLAS).
  The SPLAS is a photo-numeric rating scale ranging from 1 (none) to 5 (very severe), where higher scores indicate greater severity of static perioral lines. The investigator uses the accompanying morphed images and photo atlas to support standardized severity grading at each assessment time point.
  The outcome is expressed as the change in SPLAS score relative to baseline, reflecting changes in static perioral line severity over time.
Change in lip and perioral volume assessed by three-dimensional (3D) facial imaging | Week 6, Week 12
  Change from baseline in lip and perioral volume, assessed at Week 6 and Week 12 using three-dimensional (3D) facial imaging acquired with the VECTRA M3 imaging system (Canfield Scientific Inc., Fairfield, New Jersey, USA).
  Standardized 3D facial photographs are obtained with participants in an upright sitting position at baseline and follow-up visits. The images are analyzed using the VECTRA Software Suite®, and volume changes in the lips and perioral region are quantified by comparing baseline images with follow-up images captured at Week 6 and Week 12.
  The outcome is expressed as the change in volume relative to baseline, reflecting changes in lip and perioral volume over time.
Patient satisfaction with treatment assessed using a clinic-internal patient satisfaction questionnaire | Week 12
  Patient satisfaction with the treatment as assessed by participants using the clinic-internal questionnaire titled "Patient Satisfaction Questionnaire". The questionnaire consists of 5 questions evaluating the participant's overall satisfaction with the treatment outcome. Each item is rated on a numeric ordinal scale from 1 to 5, where lower scores indicate higher patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- YUVELL, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided